CLINICAL TRIAL: NCT02462837
Title: Myrbetriq™ (Mirabegron) to Reduce Pain and Discomfort Following Ureteral Stent Placement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient rate of accrual
Sponsor: Southern Illinois University (Other)
Collaborators: Astellas Scientific & Medical Affairs, Inc. (Industry); Sisters of the Third Order of St. Francis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MYRB-14B02
Record Dates: First submitted 2015-05-22; First posted 2015-06-04 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Urinary Bladder, Overactive; Pain; Lower Urinary Tract Symptoms
Keywords: Ureteral Stents; Pain and Discomfort; Bladder Storage Symptoms
MeSH Terms: conditions — Urinary Bladder, Overactive; Pain; Lower Urinary Tract Symptoms | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): after stent placement, patient will be given Mirabegron 50 mg, PO, once daily, for 2 weeks
  Interventions: Drug: Mirabegron
- Placebo Arm (Placebo Comparator): after stent placement, patient will be given placebo PO, once daily, for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron
  Other Names: Myrbetriq
  Arms: Treatment Arm
Drug: Placebo
  Arms: Placebo Arm

SUMMARY:
The objective of this pilot study is to assess whether Myrbetriq™ will improve post-operative ureteral pain and discomfort, reduce bladder storage symptoms and increase quality of life following ureteral stenting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Subject scheduled to undergo a ureteral stent placement for ureteral obstruction or post- ureteroscopy procedure.
3. Otherwise healthy subjects who are able and willing to participate in the study.
4. None of the planned interventions are documented in the labeled contraindications, warnings and precautions of the study drug.

Exclusion Criteria:

1. Does NOT give consent.
2. Subject is using prohibited medications which cannot be stopped safely at the screening visit. Subject is excluded if using restricted medications not meeting protocol-specified criteria:

   (i) Phytotherapy for BPH or a 5-alpha reductase inhibitor within 3 months, with persistent urinary symptoms and AUASS more than 7.

   (ii) Taken an oral alpha agonist, anticholinergic or cholinergic medication within 5 days of the first screening visit with the following exception(s): a singular dose given in ER or on the hospital floor prior to procedure, topical anticholinergic eye drops used for glaucoma or inhaled anti-cholinergic used for COPD.

   (iii) Taken tricyclic antidepressants within 2 weeks of the first screening visit.

   (iv) Taken an estrogen, androgen, or any drug producing androgen suppression, or anabolic steroids within 3 months with the following exceptions: any topical creams for local treatment.
3. Post void residual volume > 350 mL.
4. Female subject is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential is sexually active and not practicing a highly reliable method of birth control.
5. Subject has known neurogenic bladder.
6. Subject with uncontrolled chronic pain problems or on chronic pain medications.
7. Subject has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor as determined by the investigator (for female subjects confirmed by a cough provocation test).
8. Subject has an indwelling catheter or practices intermittent self-catheterization.
9. Known primary neurologic conditions such as multiple sclerosis, Parkinson's disease, diabetic neuropathy or any neurological diseases known to affect bladder function.
10. Subject has evidence of a symptomatic active urinary tract infection, chronic inflammation such as interstitial cystitis, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs, or bladder stones (which can be located in different anatomical location and can cause LUTS similar to bladder infection and pain related to their location in the bladder which could mask the treatment effect).
11. Subject who is currently under active treatment with botulinum toxin (and all other bladder paralytics) intravesically.
12. Subject has moderate to severe hepatic impairment [ALT (SGPT) or AST (SGOT) value greater than 3 times the upper limit of normal in the clinical center lab; confirmed on a second measurement].
13. Subject has severe renal impairment or End Stage Renal disease (i.e., creatinine greater than 2.0 mg/dl).
14. Subject has severe uncontrolled hypertension (defined as systolic blood pressure ≥180mmHg and /or diastolic pressure ≥ 110mmHg).
15. Subject has a clinically significant abnormal ECG in their chart or has a known history of QT prolongation or currently taking medication known to prolong the QT interval. Any patient taking Digoxin.
16. Subject has a known or suspected hypersensitivity to Mirabegron or any of the inactive ingredients.
17. Subject has a concurrent genitourinary malignancy, or active cancer (except noninvasive skin cancer) within the last 5 years prior to screening. Men with a history of prostate cancer regardless of curability are not eligible.
18. Subject has been treated with an experimental device within 30 days or received an experimental agent within the longer of 30 days or five half-lives.
19. Unable to follow protocol directions due to organic brain or psychiatric disease.
20. Intra-operative complications that require hospital admissions.
21. History of alcoholism or any other substance abuse, which, in the opinion of the investigator, would affect compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05; Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Zawahry, MD, Principal Investigator — SIUSOM - Division of Urology
Locations (1):
- SIUSOM - Division of Urology, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We consented 11 patients. Two were screen fails (SF) after consenting but prior to randomization. Two patients were early withdrawls (EW) prior to enrollment when their surgeries were moved to a non-study hospital. Of the 11 total consented, 4 dropped out resulting in a total of 7 being assigned to a treatment arm. One of the SF patients provided baseline quesionnaire date (which has been updated), the other SF and both EW did not provide any baseline information.
Groups:
- Treatment Arm: after stent placement, patient will be given Mirabegron 50 mg, PO, once daily, for 2 weeks
  Mirabegron
- Placebo Arm: after stent placement, patient will be given placebo PO, once daily, for 2 weeks
  Placebo
Period: Overall Study
Arm/Group | Treatment Arm | Placebo Arm
Started | 4 | 3
Completed | 2 | 3
Not Completed | 2 | 0
Not completed — pt developed hives | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: of the 4 patients in the treatment arm - 2 of them did not finish the study after a couple of days of enrollment due 1)hives) and 2) desire to no longer be a participant in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7
American Urological Association Symptom Score (AUASS) [Mean (Full Range); unit: units on a scale] — AUASI is a 7-item self report measure used to assess urinary urgency, frequency, and voiding symptoms. total scare depicts severity of symptoms Mild (1-7), Moderate (8-19), Severe (20-35). There is a final questions pertaining solely to quality of life that is not included in the scoring. We did not analyze any information because the enrolled number of patient who completed study was only 5. Population: of the 4 patients in the treatment arm - 2 of them did not finish the study after a couple of days of enrollment due 1)hives) and 2) desire to no longer be a participant in the study. The two who did not finish the study did complete the baseline questionnaire.
  units on a scale | 18.75 [4 to 30] | 8.67 [0 to 16] | 14.42 [0 to 30]
Patient Global Impression of Severity (PGI-S) Questionnaire [Mean (Full Range); unit: units on a scale] — This questionnaires simply asks patients to check the number that best describes how their urinary symptoms are now, compared with how it was before they had the surgery: 1. Normal 2. Mild 3. Moderate 4. Severe Population: Data provided is only for 6 patients, as 1/7 patient did not finish this questionnaire at baseline
  units on a scale
    number analyzed (Participants) | 4 | 2 | 6
    (all) | 3 [2 to 4] | 2 [1 to 3] | 2.67 [1 to 4]
Visual Analog Scale (VAS) [Mean (Full Range); unit: units on a scale] — VAS is used to score pain level of patient on a scale of 1-10.
  units on a scale | 4 [0 to 8] | 0.67 [0 to 2] | 2.57 [0 to 8]
Incontinence Symptom Severity Index (ISSI) [Mean (Full Range); unit: units on a scale] — A selfl-assessment instrument for voiding symptom severity. It assesses 8 symptom domains: emptying, urgency, urge incontinence, nocturia, daytime frequency, stress incontinence, leakage with physical activity, and pad use. absent/mild (0-6), moderate (7-16), severe (>16).
  units on a scale | 13 [3 to 19] | 4.67 [2 to 8] | 9.43 [2 to 19]

OUTCOME MEASURES:

1. Primary Outcome: Improvement From Baseline in the Incontinence Symptom Severity Index (ISSI) in the Myrbetriq™ Group at the 2 Week Follow-up Compared to Placebo Group.
Description: Incontinence symptom severity index is a self-assessment instrument for voiding symptom severity. It assesses 8 symptom domains: emptying, urgency, urge incontinence, nocturia, daytime frequency, stress incontinence, leakage with physical activity, and pad use. absent/mild (0-6), moderate (7-16), severe (>16).
Time Frame: 2 weeks
Population: Study was terminated due to insufficient rate of accrual. Only seven patients were assigned to treatment/placebo arms and two of them (both in treatment) withdrew after the first dose. Therefore, we are only left with 5 patients completing the study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 2 | 3
score on a scale | 9.5 [4 to 15] | 8 [6 to 11]

2. Primary Outcome: Improvement From Baseline in the Number Micturitions Per 24 Hours in the Myrbetriq™ Group at the 2 Week Follow-up Compared to Placebo Group.
Description: Only seven patients were enrolled and two of them withdrew after the first dose. Patients did not provide baseline micturitions. They were given a voiding diary after randomization to be conducted prior to their next follow-up visit. Therefore, improvement in the number of micturitions at 2 weeks cannot be analyzed from baseline
Time Frame: 2 weeks
Population: Study was terminated due to insufficient rate of accrual. Only seven patients were assigned to treatment/placebo arms and two of them (both in treatment) withdrew after the first dose. Therefore, we are only left with 5 patients completing the study. Patients did not provide baseline micturitions so cannot do analysis of improvemet of baseline to 2 week f/u.
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Improvement From Baseline in the Number of Incontinence Episodes in the Myrbetriq™ Group at the 2 Week Follow-up Compared to Placebo Group.
Description: Only seven patients were enrolled and two of them withdrew after the first dose. Patients did not provide baseline number of incontinence episodes. They were given a voiding diary after randomization to be conducted pror to their next follow-up visit. Therefore, improvement in the number of incontinence episodes at 2 weeks cannot be analyzed from baseline.
Time Frame: 2 weeks
Population: Study was terminated due to insufficient rate of accrual. Only seven patients were assigned to treatment/placebo arms and two of them (both in treatment) withdrew after the first dose. Therefore, we are only left with 5 patients completing the study. Patient did not provide baseline number of incidence so cannot do analysis of improvement of baseline to 2 week follow-up.
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Improvement From Baseline in the Incontinence Symptom Severity Index (ISSI) in the Myrbetriq™ Group at the 1 Week Follow-up Compared to Placebo Group.
Description: Only seven patients were enrolled and two of them withdrew after the first dose. Therefore, we are only left with 5 patients completing the study.
  Incontinence symptom severity index is a self-assessment instrument for voiding symptom severity. It assesses 8 symptom domains: emptying, urgency, urge incontinence, nocturia, daytime frequency, stress incontinence, leakage with physical activity, and pad use. absent/mild (0-6), moderate (7-16), severe (>16).
  .
Time Frame: 1 week
Population: Study was terminated due to insufficient rate of accrual. Therefore, we are only left with 5 patients completing the study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 2 | 3
score on a scale | 10 [3 to 17] | 6.67 [4 to 9]

5. Primary Outcome: Improvement From Baseline in the Number Micturitions Per 24 Hours in the Myrbetriq™ Group at the 1 Week Follow-up Compared to Placebo Group.
Description: Only seven patients were enrolled and two of them withdrew after the first dose. Therefore, we are only left with 5 patients at the one week follow-up. Patients did not provide baseline micturitions. They were given a voiding diary after randomization to be conducted prior to their next follow-up visit. Therefore, improvement in the number of micturitions at 1 week cannot be analyzed from baseline
Time Frame: 1 week
Population: Patients did not provide baseline micturitions so cannot do analysis of improvemet of baseline to 1 week f/u.
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Improvement From Baseline in the Number of Incontinence Episodes in the Myrbetriq™ Group at the 1 Week Follow-up Compared to Placebo Group.
Description: Only seven patients were enrolled and two of them withdrew after the first dose. Therefore, we are only left with 5 patients at the one week follow-up. Patients did not provide baseline number of incontinence episodes. They were given a voiding diary after randomization to be conducted pror to their next follow-up visit. Therefore, improvement in the number of incontinence episodes at 1 week cannot be analyzed from baseline.
Time Frame: 1 week
Population: Study was terminated due to insufficient rate of accrual. Patient did not provide baseline number of incidence so cannot do analysis of improvement of baseline to 1 week follow-up.
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Improvement in Pain and Discomfort Perception Using a 10 Point Visual Analog Scale for Pain Assessment (VAS) at the 1 and 2 Week Follow-up.
Description: Only seven patients were enrolled and two of them withdrew after the first dose. Therefore, we are only left with 5 patients completing the study. Visual analog scale is from 1-10 (10 being the worse possible pain).
Time Frame: 1 week, 2 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 2 | 3
score on a scale
  1 week follow/up | 4 [0 to 8] | 2.67 [0 to 6]
  2 week follow/up: number analyzed (Participants) | 2 | 2
  2 week follow/up | 4.5 [2 to 7] | 1.33 [0 to 4]

8. Secondary Outcome: Improvement From Baseline on the Patient Global Impression of Severity (PGI-S) at the 2 Week Follow-up.
Description: Only seven patients were enrolled and two of them withdrew after the fist dose. Therefore, we are only left with 5 patients completing the study. PGI-S is a four item questionnaire asking for patient enumeration of their urinary symptoms when compared to symptoms prior to surgery (1= normal, 2=mild, 3=moderate, 4=severe)
Time Frame: 2 weeks
Population: Study was terminated due to insufficient rate of accrual. Only seven patients were enrolled and two of them withdrew after the fist dose. Therefore, we are only left with 5 patients completing the study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 2 | 3
score on a scale | 2.5 [2 to 3] | 2 [1 to 3]

9. Secondary Outcome: Reduction in Pain Medicine Intake at the 2 Week Follow-up
Description: This outcome measure will be listed in 1) mean number of days that pain medications were taken
Time Frame: 2 weeks
Population: Study was terminated due to insufficient rate of accrual. Only seven patients were enrolled and two of them withdrew after the first dose. Therefore, 5 patients completed study. We are including the two early withdrawal patients in this population analysis because they did provide the pain medication log prior to withdrawal.
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 4 | 3
days | 5 [1 to 11] | 7.67 [3 to 15]

10. Secondary Outcome: Reduction in Pain Medicine Intake at the 2 Week Follow-up
Description: This outcome measure will be listed in mean number of times per day that pain medication was taken
Time Frame: 2 weeks
Population: Study was terminated due to insufficient rate of accrual. Only seven patients were enrolled and two of them withdrew after the first dose. There 5 patients completed study. We are including the two early withdrawal patients because they did provide the pain medication log prior to withdrawal.
Measure: Mean (Full Range); unit: # times per day pain medication taken
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 4 | 3
# times per day pain medication taken | 2.22 [1 to 5] | 1.4 [1 to 2]

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Description: it does not differ from the clinicaltrials.gov definitions
Arm/Group | Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=4) | Placebo Arm (N=3)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT02462837/Prot_SAP_000.pdf